CLINICAL TRIAL: NCT01635725
Title: New Bowel Preparation Scale for Measuring the Cleansing of the Colon for Colonoscopy
Brief Title: New Bowel Preparation Scale for Measuring Colon Cleanliness
Status: Completed | Type: Observational
Sponsor: Gastroenterology Services, Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: AMH 2012-08
Record Dates: First submitted 2012-07-04; First posted 2012-07-10 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Colonoscopy; Bowel Cleanliness; Bowel Rating Scale
Keywords: colonoscopy; bowel cleanliness; bowel rating scale

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this investigation is validate a new bowel preparation scale and to compare it to existing bowel preparation scales.

DETAILED DESCRIPTION:
Early studies of bowel preparations for colonoscopy relied on scales to measure the cleanliness of the colon that were not validated or sensitive to differences in preparation quality. Often these scales would simply describe the bowel preparation as adequate or inadequate based on the endoscopist's judgment of quality of the overall preparation.

An ideal bowel cleanliness scale would:

1. Produce a score that is reproducible from endoscopist to endoscopist (be validated).
2. Be easy for the endoscopist to use.
3. Produce a score that is easily converted into the poor/fair/good/excellent subjective rating scale that is often used by gastroenterologists in their colonoscopy reports.
4. Produce a score that is easily converted into the adequate/inadequate subjective rating scale that is often used by gastroenterologists in their colonoscopy reports.
5. Recognize truly outstanding preparations where 100% of the mucosa is well visualized without any cleaning required.
6. Recognize adequate preparations (the ability to visualize the mucosa), but also measure the effort required to clean the colon of residual liquid.

In 2004, a study validating the Ottawa Preparation Scale (OPS) was published (Rostom, Jolicoeur, 2004). A description of the scoring system is below:

Ottawa Preparation Scale (OPS) rating for each colon segment 4=Inadequate (Solid stool not cleared with washing and suctioning) 3=Poor (Necessary to wash and suction to obtain a reasonable view) 2=Fair (Necessary to suction liquid to adequately view segment) 1=Good (Minimal turbid fluid in segment) 0=Excellent (Mucosal detail clearly visible) Ottawa Preparation Scale (OPS) rating for the amount of fluid in the whole colon 2=Lots of fluid

1=Moderate fluid 0=Little fluid

OPS is calculated by adding the ratings of the right, transverse/descending and sigmoid/rectum colon segments and the rating for the fluid in the whole colon. The overall OPS is reported from 14 (very poor) to 0 (excellent).

Although the OPS was a major improvement over previous cleanliness scales, there were a number of significant problems with the OPS:

1. The segments rated were not easily defined by the endoscopist, especially the demarcation between the descending colon and the sigmoid colon.
2. The segment scores were based on how much cleaning was required to view the mucosa of each segment, rather than the quality of the ultimate view of the mucosa. Although it is preferred to have a colon that does not require any cleaning, the ultimate view of the mucosa is what is most important.
3. Adequate and inadequate preparations do not correlate with the OPS score. For example, if 2 segments were rated Excellent and one was rated Inadequate, then the total score would be 4 - but the colon cleansing would not be adequate for a good quality colonoscopy. If it were necessary to suction liquid from all 3 segments, then the total score would be 6 - but the colon cleansing still would be adequate and might even be excellent after cleaning.
4. The OPS suffers from a poorly designed scoring system that is not easily converted into the poor/fair/good/excellent subjective rating scale which is often used by gastroenterologists in their colonoscopy reports.
5. The OPS penalizes for liquid in the colon which does not necessarily correlate with a poorer quality view of the mucosa. Preparations given in split doses (half the night before and half the morning of the procedure) tend to be wetter because there is less time for the preparation to pass through the body. As long as the fluid is clear or easily suctioned through the colonoscopy, it does not negatively impact the ultimate of the view of the mucosa.

In 2009, a study validating the Boston Bowel Preparation Scale (BBPS) was published (Edwin, Calderwood, et al., 2009). A description of the scoring system is below:

Boston Bowel Preparation Scale (BBPS) rating for each colon segment 0=Unprepared colon segment with stool that cannot be cleared

1. Portion of mucosa in segment seen after cleaning, but other areas not seen due to retained material
2. Minor residual material after cleaning, but mucosa of segment generally well seen
3. Entire mucosa of segment well seen after washing

BBPS is calculated by adding the ratings of the right, transverse and left colon segments. The overall BBPS is reported from 0 (very poor) to 9 (excellent).

The BBPS was simpler for the endoscopist use than the OPS, it rated the ultimate cleanliness of the colon rather than the effort required to clean the colon, and the segments of the colon the endoscopist rated were anatomically easier to define. Still, there were a number of significant problems with the BBPS:

1. Adequate and inadequate preparations do not correlate with the BBPS score. For example, if the entire mucosa of 2 segments was well seen and one segment was Unprepared, then the score would be 6 - but the colon cleansing would not be adequate for a good quality colonoscopy. If it there was minor residual material after cleaning in all 3 segments, then the score would also be 6 - but the colon cleansing would be adequate for a good quality colonoscopy.
2. The BBPS suffers from poorly a designed scoring system that is not easily converted into the poor/fair/good/excellent subjective rating scale that is often used by gastroenterologists in their colonoscopy reports.
3. The BBPS does not penalize for liquid in the colon. While liquid that can be removed does not necessarily correlate with a poorer view of the mucosa, a preparation that cleans the colon well and leaves it dry would be preferred.
4. A truly outstanding colon preparation would allow 100% of the mucosa to be viewed without any cleaning. The BBPS is not very sensitive to truly outstanding preparations since it does not penalize for the effort required to clean the colon.
5. Segments of the colon which are rated 1 on the BBPS can vary greatly in cleanliness. For example, a colon where all 3 segments had 2% of the mucosa not well seen could receive a BBPS score of 3 and the preparation would be good to excellent. Another colon where each segment had 50% of the mucosa not well seen could receive a BBPS score of 3 and the preparation would be poor.

We propose to study a new bowel preparation scale that we call the "Chicago Bowel Preparation Scale" that overcomes most of the limitations of previous preparation scales.

ELIGIBILITY:
Inclusion Criteria:

* All Patients undergoing a colonoscopy in our office endoscopy suite

Exclusion Criteria:

* Patients younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients already planning to have a colonoscopy in our office endoscopy suite.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient between the PA and physician ratings of bowel cleanliness | During a Colonoscopy (about 20 min)
  The quality of the colon preparation will be graded based on the OPS, BBPS, an adequate/inadequate scale and our new CBPS. The correlation between the endoscopist's cleanliness rating and the physician assistant's cleanliness rating will be calculated using the appropriate statistical measures. These statistical measures were chosen before the study began by our statistical consultant.

SECONDARY OUTCOMES:
Correlation coefficient between the PA and physician ratings of total bowel fluid. | During a Colonoscopy (about 20 min)
  The amount of fluid present in the whole colon (excluding any fluid added to clean the mucosa) will be estimated by the physician's assistant and physician without discussing the estimate with each other. A covered suction bottle will be used to measure the actual volume of fluid suctioned. The correlation coefficient between the PA and physician ratings will be measured by statistics chosen before the study began by our statistical consultant.

CONTACTS AND LOCATIONS:
Overall Officials: David P Gerard, MD, Principal Investigator — Gastroenterology Services, Ltd.
Locations (1):
- Gastroenterology Services, Downers Grove, Illinois, United States

REFERENCES:
- [Result] Gerard DP, Foster DB, Raiser MW, Holden JL, Karrison TG. Validation of a new bowel preparation scale for measuring colon cleansing for colonoscopy: the chicago bowel preparation scale. Clin Transl Gastroenterol. 2013 Dec 5;4(12):e43. doi: 10.1038/ctg.2013.16. PMID 24304940